CLINICAL TRIAL: NCT04737174
Title: Adjunctive ES-481 for Uncontrolled Glioma-Associated Epilepsy and Assessment for Potential Anti-Tumorigenic Effect in Patients With Isocitrate Dehydrogenase 1 (IDH1) Mutant Tumors
Brief Title: ES-481 for Uncontrolled Glioma-Associated Epilepsy and Assessment for Potential Anti-Tumorigenic Effect in Patients With Isocitrate Dehydrogenase 1 (IDH1) Mutant Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of identifiable patients
Sponsor: ES Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EST-481 2020-Onco-101-HGG
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ES-481 (Experimental): Administered as 25 mg oral gelatin capsules
  Interventions: Drug: ES-481

INTERVENTIONS:
Drug: ES-481 — 28-day screening period followed by 4-week dose escalation period followed by 16-week treatment period followed by 4-week dose washout period

SUMMARY:
Phase 2A single-arm exploratory clinical study in up to 12 adult subjects aged 18 and older with primary glioma, IDH1 mutation, and uncontrolled focal-onset seizure activity to determine the potential efficacy, safety and pharmacokinetics of ES-481 as adjunctive therapy in glioma-associated epilepsy and to assess for potential anti-tumorigenic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects greater than 18 years of age
2. Subjects with brain tumour-related epilepsy
3. Subjects with a history of uncontrolled seizures (at least three focal-onset seizure per month over the last 28 days)
4. Subjects currently being treated with at least one appropriate AED
5. Subjects who have had a brain MRI performed in the last three months preceding the signing of informed consent
6. Subjects with primary brain tumour with an IDH1 mutation (to be determined during the screening period)
7. Subjects with satisfactory hematologic, renal and liver function, as assessed by the Principal Investigator
8. Subject with a Karnofsky performance scale index (KPD) of > 70%
9. An expected survival time > 6 months
10. A female subject is eligible to participate if she is not pregnant by serum pregnancy test, not breastfeeding, and at least 1 of the following conditions applies:

    1. Not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or postmenopausal (no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient)
    2. Of childbearing potential and agrees to use a highly effective method of contraception consistently during the 4-week dose escalation, 16-week treatment, and 4-week washout periods; and for at least 30 days after the last dose of study treatment
11. A male patient with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during 4-week dose escalation, 16-week treatment, and 4-week washout periods; and for at least 30 days after the last dose of study treatment and refrains from donating sperm during this period
12. Willing to participate in the study and willing to provide written signed informed consent.

Exclusion Criteria:

1. Urgent need for surgical intervention
2. Alanine aminotransferase or aspartate aminotransferase > 10 times the upper reference limit at the screening visit
3. Estimated glomerular filtration rate < 60 mL/min (calculated using the using the Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation) at the screening visit
4. Any haematological National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 Grade ≥ 3 (with the exception of alopecia) at the screening visit
5. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhoea, short bowel syndrome, and/or intestinal obstruction
6. Hypertension that cannot be reduced to normal range with antihypertensive medication (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
7. Concurrent active cancer that requires non-surgical treatment (e.g., chemotherapy, radiotherapy, adjuvant therapy)
8. History of severe cardiovascular disease: myocardial ischemia or myocardial infarction of Grade 2 or above, poorly controlled arrhythmia (including QTc interval ≥450 ms for men, ≥470 ms for women); according to New York Heart Association standards, Grade 3 or 4 cardiac insufficiency, or colour doppler ultrasound examination of the left ventricular ejection fraction < 50% as assessed at the screening visit
9. In the Investigators opinion, the subject's involvement may affect the progress of the clinical study and/or the determination of the research results, and/or considers them unsuitable for inclusion
10. Previously suffered severe cardiovascular disease: myocardial ischemia or myocardial infarction of Grade 2 or above, poorly controlled arrhythmia (including QTc interval ≥450 ms for men, ≥470 ms for women); according to New York Heart Association standards, Grade 3 or 4 cardiac insufficiency, or color doppler ultrasound examination of the left ventricular ejection fraction < 50%.
11. Investigator judges that may affect the progress of the clinical study and/or the determination of the research results, and/or considers them unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-25 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram Monitoring of epileptiform interictal and seizure discharge | Continual 24 hours
Subject Captured Seizure Activity | Continual 24 hour
  Subjects will keep daily diary of seizure activity

CONTACTS AND LOCATIONS:
Overall Officials: Terence O'Brien, MD, Principal Investigator — The Alfred Centre